CLINICAL TRIAL: NCT03341650
Title: The Effect of High Pasta vs. Low Pasta Mediterranean Diet on Weight Loss in the Treatment of Obese Patients
Brief Title: High Pasta vs. Low Pasta Diet in the Treatment of Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Parma (Other)
Responsible Party: Principal Investigator, Francesca Scazzina Ph.D., Assistant Professor, University of Parma
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SP2
Record Dates: First submitted 2017-11-07; First posted 2017-11-14 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2017-11

CONDITIONS: Diet Therapy
Keywords: Mediterranean Diet; BMI; weight loss; pasta; obesity
MeSH Terms: conditions — Weight Loss; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Pasta (Experimental): Habitual pasta consumption equal or higher than 5 times/week.
  Interventions: Behavioral: High Pasta
- Low Pasta (Experimental): Habitual pasta consumption equal or lower than 3 times/week.
  Interventions: Behavioral: Low Pasta

INTERVENTIONS:
Behavioral: High Pasta — Participants received a personalised diet program considering their food preferences and eating behaviour, based on the Italian guidelines for a healthy and Mediterranean diet and were encouraged to maintain their habitual consumption of pasta (at least 5 times/week). To encourage participants to prepare healthy meals by using high-quality ingredients, participants were provided with a recipe book and dietary guidelines and recommendations.
  Arms: High Pasta
Behavioral: Low Pasta — Participants received a personalised diet program considering their food preferences and eating behaviour, based on the Italian guidelines for a healthy and Mediterranean diet and were encouraged to maintain their habitual consumption of pasta (no more than 3 times/week). To encourage participants to prepare healthy meals by using high-quality ingredients, participants were provided with a recipe book and dietary guidelines and recommendations.
  Arms: Low Pasta

SUMMARY:
To the best of our knowledge, the effect of pasta consumption within a hypocaloric Mediterranean diet has only been scarcely explored yet. Therefore, a two-parallel group dietary intervention was carried out to investigate if pasta consumption could affect the BMI change in obese patients. The primary outcome was the loss of at leat 8% of the initial body weight in the first 6 months. Anthropometric and body composition (from bioelectrical impedance analysis - BIA-) measures were collected every month for the first 6 months and after 1 year. In addition, dietary information was collected at baseline and after 3, 6 and 12 months through a 7-day carbohydrate food record and a 24-h food recall. Blood samples were collected at baseline and at 6 and 12 months to assess: glucose, insulin, Homeostatic model assessment for insulin resistant (HOMA-IR) index, total cholesterol, low-density lipoprotein, high-density lipoprotein, and uric acid. Furthermore, the perceived quality of life was investigated through the 36-items short form health survey (SF36) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 30-45 kg/m2
* healthy subjects
* regular meal consumption
* no celiac disease
* no menopause woman

Exclusion Criteria:

* with a BMI <30 or >45 kg/m2
* having diabetes, hepatic or kidney diseases
* having an eating disorder
* having celiac disease
* menopause woman

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2015-11-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline Body weight at 6 months | baseline, 6 months
  Measured in kg according to the standard procedure

SECONDARY OUTCOMES:
Change from baseline Body weight at 3 months | baseline, 3 months
  Measured in kg according to the standard procedure
Change from baseline Body weight at 12 months | baseline, 12 months
  Measured in kg according to the standard procedure
BMI | baseline, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months, 12 months
  Calculated as body weight in kilograms divided by the square of the height in meters
Waist circumference | baseline, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months, 12 months
  Measured in cm according to the standard procedure
Free Fat Mass | baseline, 3 months, 6 months, 12 months
  Estimated by bioelectrical impedance analysis in kg and in %
Fat Mass | baseline, 3 months, 6 months, 12 months
  Estimated by bioelectrical impedance analysis in kg and in %
Basal Metabolic Rate | baseline, 3 months, 6 months, 12 months
  Estimated by bioelectrical impedance analysis in kcal/day
Glucose | baseline, 6 months, 12 months
  mg/dL in fasting condition
Insulin | baseline, 6 months, 12 months
  microU/mL in fasting condition
HOMA-IR index | baseline, 6 months, 12 months
  calculated from glucose and insulin in fasting condition
Total cholesterol | baseline, 6 months, 12 months
  mg/dL in fasting condition
HDL cholesterol | baseline, 6 months, 12 months
  mg/dL in fasting condition
LDL cholesterol | baseline, 6 months, 12 months
  mg/dL in fasting condition
Triglycerides | baseline, 6 months, 12 months
  mg/dL in fasting condition
Uric Acid | baseline, 6 months, 12 months
  mg/dL in fasting condition
Energy intake | baseline, 3 months, 6 months, 12 months
  assessed by a 24-h dietary recall as kcal/day
Nutrient intakes | baseline, 3 months, 6 months, 12 months
  assessed by a 24-h dietary recall as g/day
Carbohydrate-based food intakes | baseline, 3 months, 6 months, 12 months
  assessed by a 7-day food diary as times/week
Perceived Quality of Life | baseline, 3 months, 6 months, 12 months
  assessed by the SF36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Dall'Aglio, MD, Study Director — University of Parma
Locations (1):
- Department of Food and Drug, University of Parma, Parma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rosi A, Tesan M, Cremonini A, Biasini B, Bicchieri L, Cossu M, Brighenti F, Dall'Aglio E, Scazzina F. Body weight of individuals with obesity decreases after a 6-month high pasta or low pasta Mediterranean diet weight-loss intervention. Nutr Metab Cardiovasc Dis. 2020 Jun 9;30(6):984-995. doi: 10.1016/j.numecd.2020.02.013. Epub 2020 Feb 24. PMID 32402585